CLINICAL TRIAL: NCT07269197
Title: The Association of Sodium-Glucose Cotransporter 2 Inhibitors Therapy With Elastographic and Molecular Markers of Liver Injury in Patients With Type 2 Diabetes Mellitus
Brief Title: Association of SGLT2 Inhibitors Therapy With Elastographic and Molecular Markers of Liver Injury in Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Josip Juraj Strossmayer University of Osijek (Other)
Responsible Party: Principal Investigator, Farah Khaznadar, Principal Investigator, Josip Juraj Strossmayer University of Osijek
Other Study IDs: 2158-61-46-23-122
Record Dates: First submitted 2025-11-17; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Diabetes Mellitus, Type 2
Keywords: elastography; UGAP; MASLD; SGLT2 inhibitor; fatty liver; empagliflozin; dapagliflozin; Diabetes mellitus type 2
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Diabetes Mellitus, Type 2; Fatty Liver | interventions — dapagliflozin; empagliflozin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Sodium Glucose Co-transporter 2 (SGLT2) Inhibitor — In patients with T2DM initiating therapy with a SGLT2 inhibitor, the effects on the liver have been assessed.
  Other Names: Dapagliflozin; Empagliflozin; Jardiance; Forxiga

SUMMARY:
Metabolic dysfunction-associated steatotic liver disease (MASLD), a condition where fat builds up in the liver, is common in patients with type 2 diabetes. Sodium-glucose cotransporter 2 (SGLT2) inhibitors may help improve liver health, but their effects on liver stiffness and fat are not yet well understood. This study aims to clarify these effects.

Therefore, the aims of this study are:

1. Measurement of liver stiffness and liver steatosis using novel ultrasound-based methods before initiating SGLT2 inhibitor therapy and 6 months after starting therapy.
2. Assessment of blood biomarkers that may indicate liver injury, increased fat accumulation, and cellular dysfunction before initiating SGLT2 inhibitor therapy and 6 months after starting therapy.
3. Evaluation of the relationship between biomarkers and ultrasound findings before the introduction of SGLT2 inhibitors and 6 months after the start of therapy.

DETAILED DESCRIPTION:
Metabolic dysfunction-associated steatotic liver disease (MASLD) is highly prevalent among patients with type 2 diabetes mellitus (T2DM), yet targeted therapeutic strategies remain limited. Sodium-glucose cotransporter 2 (SGLT2) inhibitors have demonstrated favorable metabolic and potential hepatoprotective effects, however, their impact on liver stiffness and steatosis has not been fully characterized.

This study was conducted to assess the effects of SGLT2 inhibitor therapy on non-invasive elastographic parameters and markers of liver injury in patients with T2DM. Liver stiffness was assessed using two-dimensional shear wave elastography (2D-SWE) and liver steatosis using ultrasound-guided attenuation parameter (UGAP), at baseline and after 6 months of treatment.

Comprehensive biochemical analysis was performed, including glucose, HbA1c, hematologic parameters, and standard liver function markers (AST, ALT, GGT, ALP, coagulation profile, albumin, total proteins, total and conjugated bilirubin, and lipid profile). Additionally, serum concentrations of key regulators of lipogenesis: Sterol Regulatory Element-Binding Protein 1 (SREBP1), Peroxisome Proliferator-Activated Receptor alpha (PPAR-α), Peroxisome Proliferator-Activated Receptor gamma (PPAR-γ), and Microsomal Triglyceride Transfer Protein (MTTP), were assessed at both time points.

The analysis aims to determine whether SGLT2 inhibitor therapy is associated with measurable improvements in liver stiffness, steatosis, and molecular markers of hepatic metabolic dysfunction, as well as to explore correlations between elastographic findings and circulating biomarkers. The results are expected to inform future research on the utility of these markers for diagnosing and monitoring MASLD and to support the potential expansion of therapeutic indications for SGLT2 inhibitors.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent, information for the participants and questionnaire
2. Patients that are 18 years of age or older
3. Diagnosis of type 2 diabetes mellitus
4. Patients being treated with an SGLT2 inhibitor for the first time
5. Patients who have been on stable antihyperglycemic therapy for 90 days (3 months) before enrollment in the study

Exclusion Criteria:

1. Patients taking drugs that are extremely hepatotoxic, i.e., require additional monitoring of liver function during therapy (e.g., chemotherapeutic agents, biological therapy)
2. Patients taking drugs which cause drug-induced fatty liver disease (DIFLD): amiodarone, tamoxifen, methotrexate, 5-Fluorouracil, irinotecan, l-asparaginase, valproate, tetracycline, nucleoside reverse transcriptase inhibitors (NRTIs such as lamivudine, tenofovir, zidovudine etc.)
3. Patients with liver cancer, hemochromatosis, primary biliary cholangitis (PBC), primary sclerosing cholangitis (PSC), hepatitis C virus (HCV), hepatitis B virus (HBV), liver cirrhosis or autoimmune hepatitis.
4. Patients who are alcohol addicted, i.e., consume more than two alcoholic beverages per day (for women) or more than three alcoholic beverages per day (for men)
5. Mentally ill patients who are incapable of making their own independent decisions and have a legal custodian
6. Pregnant women and nursing mothers
7. Patients who are on insulin therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Type 2 Diabetes Mellitus who have been prescribed SGLT2 inhibitor for the first time in eastern Croatia region.
Sampling Method: Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2024-03-22 (Actual); Primary Completion 2025-10-10 (Actual); Study Completion 2025-10-10 (Actual)

PRIMARY OUTCOMES:
Change in liver fibrosis (kPa) | Baseline, after 6 months
  Liver fibrosis is assessed using the two-dimensional shear wave elastography (2D-SWE)
Change in liver steatosis (dB/cm/MHz) | Baseline, after 6 months
  Liver steatosis is assessed using the ultrasound-guided attenuation parameter (UGAP).
Change in glucose levels (mmol/L) | Baseline, after 6 months
  Assessment via biochemical analyses
Change in HbA1c (%) | Baseline, after 6 months
  Assessment via biochemical analyses
Change in HbA1c (mmol/mol) | Baseline, after 6 months
  Assessment via biochemical analyses
Change in enzyme activity (U/L) of AST, ALT, GGT, ALP | Baseline, after 6 months
  Assessment via biochemical analyses
Change in Prothrombin Time ratio and change in activated Partial Thromboplastin Time ratio | Baseline, after 6 months
  Assessment via biochemical analyses
Change in Prothrombin Time-INR | Baseline, after 6 months
  Assessment via biochemical analyses
Change in fibrinogen activity (g/L) | Baseline, after 6 months
  Assessment via biochemical analyses
Change in Thrombin Time (s) and change in activated Partial Thromboplastin Time (s) | Baseline, after 6 months
  Assessment via biochemical analyses
Change in concentration (g/L) of albumins and total proteins | Baseline, after 6 months
  Assessment via biochemical analyses
Change in concentration (µmol/L) of total bilirubin and conjugated bilirubin | Baseline, after 6 months
  Assessment via biochemical analyses
Change in concentration (mmol/L) of total cholesterol, LDL cholesterol, HDL cholesterol and triglycerides | Baseline, after 6 months
  Assessment via biochemical analyses
Change in in White Blood Cell (WBC) Count (x 10^9/L) and Platelet Count (x 10^9/L) | Baseline, after 6 months
  Assessment via biochemical analyses
Change in Red Blood Cell (RBC) Count (x 10^12/L) | Baseline, after 6 months
  Assessment via biochemical analyses
Change in Hemoglobin concentration (g/L) | Baseline, after 6 months
  Assessment via biochemical analyses
Change in Hematocrit ratio (L/L) | Baseline, after 6 months
  Assessment via biochemical analyses
Change in concentration (ng/L) of SREBP-1, PPAR alpha, PPAR gamma and MTTP | Baseline, after 6 months
  Assessment via ELISA

SECONDARY OUTCOMES:
Questionnaire on lifestyle and dietary habits | Baseline, after 6 months
  Responses from a study-specific questionnaire including investigator-measured variables (weight [kg], height [cm], BMI [kg/m^2], blood pressure [mmHg], waist circumference [cm]) and patient-reported items (education, medical conditions, medications and side effects, recent antibiotic use, pregnancy/breastfeeding, supplement use). Lifestyle behaviors include alcohol intake, tobacco use, and physical activity (1 = never to 4 = very often). Dietary habits include frequency of consuming vegetables, fruits, meat, dairy, and high-calorie/junk foods (1 = almost never to 4 = very often). The questionnaire does not generate a composite or total score. Each variable will be analyzed individually as categorical, continuous, or ordinal data, depending on the question type.

CONTACTS AND LOCATIONS:
Overall Officials: Martina Smolić, MD, PhD, Study Director — Faculty of dental medicine and health Osijek, Josip Juraj Strossmayer University Osijek, 31000 Osijek, Croatia
Locations (1):
- Health Center Osijek-Baranja County, Osijek, Croatia

IPD SHARING:
Plan to Share IPD: No